CLINICAL TRIAL: NCT02746484
Title: ABILITY - TelerehABILITation. TechnologY-enhanced Multi-domain at Home Continuum of Care Program for People With Cognitive Impairment.
Brief Title: ABILITY - TelerehABILITation: TechnologY-enhanced Multi-domain at Home Continuum of Care Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FdG_AD_02
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cognitive Impairments; Dementia; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Ability platform program (Experimental): Multi-domain at home rehabilitation program delivered through the Ability platform.
  Interventions: Other: Ability platform program
- Usual care program (Active Comparator): Usual care at home program (paper and pencil cognitive activities; promotion of physical activity according to healthcare professional's advice)
  Interventions: Other: Usual care program

INTERVENTIONS:
Other: Ability platform program — The Ability program is an at home participant-tailored and technology-enhanced platform a) delivering tablet-based intensive (five days/a week for six weeks) motor and cognitive activities; b) monitoring from remote vital and physical health parameters (i.e., weight, Heart Rate, O2 saturation, daily steps, sleep activity).
  Arms: Ability platform program
Other: Usual care program — Usual care at home program (paper and pencil cognitive activities; promotion of physical activity according to healthcare professional's advice)
  Arms: Usual care program

SUMMARY:
The Ability research project, funded in Italy within the Smart Cities and Smart Communities funding program (MInistry of University and Research, Operational Regional Programme, Lombardy, Axis 1, Operational Regional Programme - European Funding for Regional Development 2007-2013), aims at developing and testing the efficacy and the impact of a Personal Smart Health Community able to provide innovative trajectories for people with cognitive impairment, putting them at the core of a continuous and intertwining treatment and support from both formal (e.g. physicians) and informal (e.g. near relatives) caregivers, with special focus on home-based care.

Within this framework of the Ability project the investigators test the efficacy of the home-based motor-cognitive rehabilitation program delivered with two different approaches: the Ability platform versus the usual care program

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as mild AD or MCI due to AD (Albert et al, 2011) according to DSM 5 diagnostic criteria (American Psychiatric Association, 2013);
* MMSE score >18
* school attendance (≥ 3 years).

Exclusion Criteria:

* dysmetria;
* serious deficits in visual acuity, acoustic perception, and in routine communication skills.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
activities of daily living | change from baseline after 8 weeks (aMCI/AD subjects)
  Activities of Daily Living Inventory (ADCS/ADL)
behavioral symptoms | change from baseline after 8 weeks (aMCI/AD subjects)
  Neuropsychiatric Inventory (NPI) score
cognitive domain (long-term memory) | change from baseline after 8 weeks (aMCI/AD subjects)
  Free and Cued Selective Recall Test (FCSRT) score
cognitive domain (language) | change from baseline after 8 weeks (aMCI/AD subjects)
  Fluency score
cognitive domain (frontal-executive functions) | change from baseline after 8 weeks (aMCI/AD subjects)
  Trail Making Test (TMT) score
quality of life | change from baseline after 8 weeks (aMCI/AD subjects)
  Dementia Quality of Life (D-QoL) Instrument
coping strategies | change from baseline after 8 weeks (aMCI/AD subjects)
  Coping Orientation for Problems Experienced - Brief Version (Brief COPE)
global cognitive level | change from baseline after 12 months (aMCI/AD subjects)
  Montreal Cognitive Asssessment (MoCA) score

SECONDARY OUTCOMES:
activities of daily living | change from baseline after 12 months (aMCI/AD subjects)
  Activities of Daily Living Inventory (ADCS/ADL)
conversion rate MCI versus AD | change from baseline after 12 months (aMCI subjects)
  conversion rate score
cognitive domain - long term memory | change from baseline after 12 months (aMCI/AD subjects)
  Free and Cued Selective Recall Test (FCSRT) score
cognitive domain - language | change from baseline after 12 months (aMCI/AD subjects)
  Fluency score
cognitive domain - frontal executive functions | change from baseline after 12 months
  Trail Making Test (TMT) score
quality of life | change from baseline after 12 months
  Dementia Quality of Life (D-QoL) Instrument
coping strategies | change from baseline after 12 months
  Coping Orientation for Problems Experienced - Brief Version (Brief COPE)
caregiver quality of life | change from baseline after 8 weeks and after 12 months
  Psychological Well-Being (PWB) scale
caregiver coping strategies | change from baseline after 8 weeks and after 12 months
  Coping Orientation for Problems Experienced - Brief Version (Brief COPE)
caregiver burden | change from baseline after 8 weeks and after 12 months
  Caregiver Burden Inventory (CBI)
caregiver affect | change from baseline after 8 weeks and after 12 months
  Positive and Negative Affect Schedule (PANAS)

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Derived] Realdon O, Rossetto F, Nalin M, Baroni I, Cabinio M, Fioravanti R, Saibene FL, Alberoni M, Mantovani F, Romano M, Nemni R, Baglio F. Technology-enhanced multi-domain at home continuum of care program with respect to usual care for people with cognitive impairment: the Ability-TelerehABILITation study protocol for a randomized controlled trial. BMC Psychiatry. 2016 Nov 25;16(1):425. doi: 10.1186/s12888-016-1132-y. PMID 27887597